CLINICAL TRIAL: NCT01878630
Title: Telemedical Interventional Management in Heart Failure II
Acronym: TIM-HF2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University of Leipzig (Other)
Responsible Party: Principal Investigator, Friedrich Koehler, Prof. Dr. Friedrich Koehler, MD, Senior Physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13KQ0904B
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; CHF

STUDY DESIGN:
Intervention Model Description: Remote patient management with telemedical devices (ECG, scale, blood-pressure device)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Patient Management (Experimental): intervention group
  Interventions: Device: Remote Patient Management
- Usual Care (Active Comparator): control group
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Remote Patient Management — Guideline-based care in heart failure including at least 5 scheduled doctor's visits within 12 months (GP and specialist) plus devices for Remote Patient Management at patient site for daily monitoring of ECG, weight, blood pressure, self-report of health status:
  * weighing scale (Seca 861 with bluetooth, seca gmbh & co. kg.)
  * blood pressure device (UA767PBT with bluetooth, A&D Ltd.)
  * ECG-eventrecorder (PhysioMem® PM 1000, getemed Medizin- und Informationstechnik AG)
  * patient-communication platform (Physio-Gate® PG 1000, getemed Medizin- und Informationstechnik AG)
  * help call device (DORO Easy 510/ Doro HandlePlus 334gsm, doro AB)
  at center site:
  - electronic patient record (eHealth connect 2.0, T-Systems International)
  Other Names: R&D project "Fontane"
  Arms: Remote Patient Management
Other: Usual Care — Guideline-based care in heart failure including at least 5 scheduled doctor's visits within 12 months (GP and specialist)
  Arms: Usual Care

SUMMARY:
Superiority of additional Remote Patient Management (RPM) in patients with chronic heart failure (CHF) in comparison to usual care in terms of, e.g.:

* days lost due to unplanned cardiovascular hospitalization or death
* all-cause mortality
* cardiovascular mortality
* quality of life

DETAILED DESCRIPTION:
The clinical trial assesses 1,500 patients over a period of 12 months each (2013 until 2015). All participants will continue to receive usual care from their general practitioner and specialist. All patients will be examined at the beginning of the study and will undergo a check-up every 3 months. 750 of the patients will be randomly allocated to receive devices for Remote Patient Management (RPM) which will measure various parameters on a daily basis (e.g. weight, blood pressure, heart rate). The devices are mobile and can be used at home or elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure New York Heart Association (NYHA) class II or III
* echocardiographically determined left ventricular ejection fraction (LVEF) ≤45% or >45% + minimum 1 diuretic in permanent medicinal therapy
* hospitalization due to decompensated HF within the last 12months before randomization
* informed consent
* Depression score PHQ-9: <10

Exclusion Criteria:

* hospitalization within the last 7 days before randomization
* implanted cardiac assist system
* acute coronary syndrome within the last 7 days before randomization
* high urgent listed for heart transplantation (HTx)
* planned revascularization, Transcatheter Aortic Valve Implantation (TAVI), MitraClip and/or Cardiac Resynchronization Therapy (CRT)-implantation within the last 3 months before randomization
* revascularization and/or CRT-implantation within 28 days before randomization
* known alcohol or drug abuse
* terminal renal insufficiency with hemodialysis
* impairment or unwillingness to use the telemonitoring equipment (e.g. dementia, impaired self-determination, lacking ability to communicate)
* existence of any disease reducing life expectancy to less than 1 year
* age <18 years
* pregnancy
* participation in other treatment studies or remote patient management programmes (register studies possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1571 (Actual)
Dates: Start 2013-08-08; Primary Completion 2017-05-12 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Percentage of days lost due to unplanned cardiovascular (CV) hospitalisation or due to death for any reason during the individual patient follow-up time. | 12 months/ individual-patient follow-up time.
  The primary outcome analysis will be performed on the FAS using the adjudicated data and sensitivity analyses will be performed on a) the PP data set, and b) on the FAS censoring all data at day 365.

SECONDARY OUTCOMES:
All-cause mortality during the individual patient follow-up time. | individual patient follow-up time (+28 days of the final visit to a maximum 393 days)
  All-cause and cardiovascular mortality will be calculated as: The individual follow-up time as calculated for the primary outcome + 28 days for all patients to a maximum of 393 days.
Percentage of days lost due to unplanned cardiovascular hospitalisations during the individual patient follow-up time. | 12 months/ individual follow-up time
Percentage of days lost due to unplanned HF-hospitalisations during the individual patient follow-up time | 12 months/ individual follow-up time
Change in MLHFQ-questionnaire overall score between baseline and 365 days | 12 months/ individual follow-up time
  The change in MLHFQ (Minnesota Living with Heart Failure Questionnaire) scores will be analysed using an analysis of covariance and the corresponding estimates with 95% confidence intervals and p-values will be provided.
Change in levels of NT-proBNP and of MR-proADM between baseline and 365 days. | 12 months/ individual follow-up time
  The change in NT-proBNP and of MR-proADM levels will be analysed using an analysis of covariance and the corresponding estimates with 95% confidence intervals and p-values will be provided

OTHER OUTCOMES:
Change in Quality of life (QoL), depression and self-care behaviour between baseline and 365 days. | 12 months (baseline and final visit)
  QoL measured by European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L), depression by PHQ-9D and self-care behaviour by European Heart Failure Self-care Behaviour Scale (EHFScBS-9)
Change from baseline in biomarkers (MR-proADM, NT-proBNP, MR-proANP, PCT) stratified by LVEF (>45 vs ≤ 45) at 365 days. | 12 months (baseline and final visit)
Unplanned cardiovascular hospitalisations and cardiovascular mortality. | individual patient follow-up time (+28 days of the final visit to a maximum 393 days)
  Analysed as a recurrent event analysis
Unplanned cardiovascular hospitalisations and all-cause mortality. | individual patient follow-up time (+28 days of the final visit to a maximum 393 days)
  Analysed as a recurrent event analysis
Unplanned heart failure hospitalisations and cardiovascular mortality. | individual patient follow-up time (+28 days of the final visit to a maximum 393 days)
  Analysed as a recurrent event analysis
Unplanned heart failure hospitalisations and all-cause mortality. | 12 month
  analysed as a recurrent event analysis
Cost-utility Analysis. | 12 month/individual follow-up time
  QALY-analysis using EQ-5D-3L
Rate of unplanned cardiovascular hospitalisations after a first cardiovascular hospitalisation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Koehler, Prof. Dr., Principal Investigator — Charité - Universitaetsmedizin Berlin
Locations (108):
- Germany (108):
  - Klinikum St. Marien Amberg - Medizinische Klinik I, Amberg
  - GLG Fachklinik Wolletzsee GmbH, Angermünde
  - Klinik Ernst von Bergmann Bad Belzig gGmbH - Zentrum für Innere Medizin/Kardiologie, Bad Belzig
  - Oder-Spree-Krankenhaus Beeskow GmbH, Beeskow
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Bundeswehr Krankenhaus, Berlin
  - Cardio Centrum Berlin GmbH, Berlin
  - DRK Kliniken Berlin-Köpenick, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe Klinik für Anthroposophische Medizin, Berlin
  - Gemeinschaftspraxis am Bayerischen Platz, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - HELIOS Klinikum Emil von Behring - HELIOS Kliniken GmbH, Berlin
  - Herzpraxis Berlin, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - Kardiologie Weissensee, Berlin
  - Kardiologische Praxis im Spreebogen, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Kranoldpraxis, Berlin
  - Martin-Luther Krankenhaus, Berlin
  - MVZ Treffpunkt Geißenweide GmbH, Berlin
  - Polikum Institut GmbH Polikum Friede, Berlin
  - Praxis am Dachsbau, Berlin
  - Praxis Claus, Berlin
  - Praxis Dres. Weinrich, Berlin
  - Praxis Frank, Berlin
  - Praxis Pinkwart, Berlin
  - Praxis Roeder, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Vivantes Klinikum Hellersdorf, Berlin
  - Vivantes MVZ Wedding, Berlin
  - Ärzte Schönhauser Berlin e.V., Berlin
  - Brandenburgklinik Berlin-Brandenburg GmbH, Bernau
  - Immanuel Klinikum Bernau, Herzzentrum Brandenburg, Bernau
  - Kardiologische Praxis Gola, Bernau
  - Gemeinschaftspraxis Hampel/Janoske, Bitterfeld-Wolfen
  - Gesundheitszentrum Bitterfeld/Wolfen gGmbH - Zentrum für Innere Medizin/Herzkatheterlabor, Bitterfeld-Wolfen
  - Städtisches Klinikum Brandenburg/Havel, Brandenburg/Havel
  - Herz - und Gefäßzentrum am Neumarkt, Celle
  - Medizinisches Beratungs- und Therapie-Zentrum Chemnitz GmbH, Chemnitz
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Klinikum Lippe - Kardiologie, Detmold
  - Cardiologicum Dresden & Pirna, Dresden
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Kreisklinik Ebersberg gGmbH, Ebersberg
  - Klinikum Barnim GmbH, Werner Forßmann Krankenhaus, Eberswalde
  - Praxis Hagenow, Elsterwerda
  - Klinikum der Johann-Wolfgang Goethe-Universität, Frankfurt am Main
  - Praxis Langel, Gera
  - Kardiologische Praxis Dr. Wehr, Gerlingen
  - Cardiocampus - Kardiologische Gemeinschaftspraxis, Gifhorn
  - Praxis Dr. med. Frank Warzok, Gotha
  - Praxis Karsten Müller, Gräfenhainichen
  - Praxis Dr. med Karsten Müller, Gräfenhainichen
  - Universitätsklinikum Halle (Saale), Halle
  - Albertinen-Krankenhaus/Albertinen-Haus gemeinnützige GmbH, Hamburg
  - Medizinische Hochschule Hannover -Klinik für Kardiologie und Angiologie/ Zentrum Innere Medizin, Hanover
  - Universitätsklinikum Jena, Jena
  - Kardiologie im Praxishaus, Kleinmachnow
  - Klinikum Dahme-Spreewald GmbH/Achenbach-Krankenhaus, Königs Wusterhausen
  - HELIOS Klinik Köthen - Klinik für Innere Medizin, Schwerpunkt Kardiologie, Internistische Intensivmedizin, Köthen
  - Asklepios Klinik Langen, Langen
  - Universitätsklinikum Leipzig - Abteilung Kardiologie & Angiologie, Leipzig
  - MVZ Lübbenau GmbH, Lubnjow
  - Cardio Centrum Ludwigsburg Bietigheim, Ludwigsburg
  - Kardiologische Gemeinschaftspraxis Dr. med. Bartels, Dr. med. Kausche, Dr. med. Meltendorf, Magdeburg
  - Dietrich Bonhoeffer Klinikum - Klinik für Innere Medizin 4, Malchin
  - Praxis Horn, Manschnow
  - Praxis Dr. med. Dieter Böhm, Marbach
  - Praxis Dr. Jens Taggeselle, Markkleeberg
  - Carl-von-Basedow-Klinikum Saalekreis gGmbH, Klinikum Merseburg, Merseburg
  - Kardiologische Praxis Dr. Rheinert, Merzig
  - Kardiologie Mühldorf am Inn, Mühldorf
  - Kardiologische Praxis Nauen, Nauen
  - Dietrich Bonhoeffer Klinikum, Neubrandenburg
  - Ruppiner Kliniken GmbH, Neuruppin
  - Kardiologische Praxis Dr. H.P. Mieg, Oranienburg
  - Praxis Donaubauer, Oschatz
  - Internist; Facharzt für Innere Medizin, Pasewalk
  - Kreiskrankenhaus Prignitz gGmbH, Perleberg
  - Cardiologicum, Pirna
  - St. Josefs-Krankenhaus Potsdam-Sanssouci, Potsdam
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
  - Poliklinik Ernst von Bergmann GmbH, Potsdam
  - Praxis Ehlert, Pritzwalk
  - Gemeinschaftspraxis Dres. Stenzel/Ebert/Otto, Riesa
  - Kardiologische Praxis Dr. Placke, Rostock
  - Facharzt-Zentrum Pneumologie und Kardiologie, Rüdersdorf
  - Klinik am See/REHA-Fachklinik für Innere Medizin, Rüdersdorf
  - Praxis für Kardiologie, Saalfeld
  - Thüringen-Kliniken "Georgius Agricola", Saalfeld
  - Bergarbeiter-Krankenhaus Schneeberg GmbH - Innere Medizin/Kardiologie, Schneeberg
  - Kliniken des Landkreises Lörrach GmbH, KKH Schopfheim, Schopfheim
  - Asklepios Klinikum Uckermark GmbH - Asklepios Kliniken GmbH, Schwedt
  - Praxis für Kardiologie, Seelow
  - Praxisklinik Herz und Gefäße - ZWEIGPRAXIS Brandenburg, Senftenberg
  - Johanniter-Krankenhaus Genthin-Stendal GmbH, Stendal
  - Internistische Gemeinschaftspraxis Steiner Thor, Straubing
  - Klinikum St. Elisabeth Straubing GmbH, Straubing
  - Internistische Praxis am Landsberger Tor, Strausberg
  - Kardiologische Facharztpraxis Dr. med. Heike Olthoff, Strausberg
  - Robert Bosch Krankenhaus Stuttgart, Stuttgart
  - Sana-Kliniken Berlin-Brandenburg GmbH, Templin
  - Kardiologische Gemeinschaftspraxis Wittenberg, Wittenberg
  - Praxis Stiller, Wittstock
  - Ambulantes Herz-Kreislauf Zentrum Wolfsburg, Wolfsburg
  - Universitätsklinikum Würzburg, Würzburg
  - Praxis Lägel, Zeuthen

REFERENCES:
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, de Brouwer S, Perrin E, Baumann G, Gelbrich G, Boll H, Honold M, Koehler K, Kirwan BA, Anker SD. Telemedicine in heart failure: pre-specified and exploratory subgroup analyses from the TIM-HF trial. Int J Cardiol. 2012 Nov 29;161(3):143-50. doi: 10.1016/j.ijcard.2011.09.007. Epub 2011 Oct 8. PMID 21982700
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Baumann G, Honold M, Koehler K, Gelbrich G, Kirwan BA, Anker SD; Telemedical Interventional Monitoring in Heart Failure Investigators. Impact of remote telemedical management on mortality and hospitalizations in ambulatory patients with chronic heart failure: the telemedical interventional monitoring in heart failure study. Circulation. 2011 May 3;123(17):1873-80. doi: 10.1161/CIRCULATIONAHA.111.018473. Epub 2011 Mar 28. PMID 21444883
- [Background] Anker SD, Koehler F, Abraham WT. Telemedicine and remote management of patients with heart failure. Lancet. 2011 Aug 20;378(9792):731-9. doi: 10.1016/S0140-6736(11)61229-4. PMID 21856487
- [Background] Cowie MR, Bax J, Bruining N, Cleland JG, Koehler F, Malik M, Pinto F, van der Velde E, Vardas P. e-Health: a position statement of the European Society of Cardiology. Eur Heart J. 2016 Jan 1;37(1):63-6. doi: 10.1093/eurheartj/ehv416. Epub 2015 Aug 24. No abstract available. PMID 26303835
- [Derived] Kerwagen F, Stork S, Koehler K, Vettorazzi E, Bauser M, Zernikow J, Barzen G, Hiddemann M, Groschel J, Gross M, Melzer C, Stangl K, Hindricks G, Koehler F, Winkler S, Spethmann S. Rurality, travel distance, and effectiveness of remote patient management in patients with heart failure in the TIM-HF2 trial in Germany: a pre-specified analysis of an open-label, randomised controlled trial. Lancet Reg Health Eur. 2025 May 18;54:101321. doi: 10.1016/j.lanepe.2025.101321. eCollection 2025 Jul. PMID 40672055
- [Derived] Koehler F, Koehler J, Bramlage P, Vettorazzi E, Wegscheider K, Lezius S, Spethmann S, Iakoubov R, Vijayan A, Winkler S, Melzer C, Schutt K, Dessapt-Baradez C, Paar WD, Koehler K, Muller-Wieland D. Impact of telemedical management on hospitalization and mortality in heart failure patients with diabetes: a post-hoc subgroup analysis of the TIM-HF2 trial. Cardiovasc Diabetol. 2024 Jun 12;23(1):198. doi: 10.1186/s12933-024-02285-0. PMID 38867198
- [Derived] Kerwagen F, Koehler K, Vettorazzi E, Stangl V, Koehler M, Halle M, Koehler F, Stork S. Remote patient management of heart failure across the ejection fraction spectrum: A pre-specified analysis of the TIM-HF2 trial. Eur J Heart Fail. 2023 Sep;25(9):1671-1681. doi: 10.1002/ejhf.2948. Epub 2023 Jul 31. PMID 37368507
- [Derived] Deckwart O, Koehler K, Lezius S, Prescher S, Koehler F, Winkler S. Effects of remote patient management on self-care behaviour in heart failure patients: results from the randomized TIM-HF2 trial. Eur J Cardiovasc Nurs. 2023 Dec 14;22(8):786-794. doi: 10.1093/eurjcn/zvad019. PMID 36752782
- [Derived] Prescher S, Winkler S, Riehle L, Hiddemann M, Moeller V, Collins C, Deckwart O, Spethmann S. Patient reported experience and adherence to remote patient management in chronic heart failure patients: a posthoc analysis of the TIM-HF2 trial. Eur J Cardiovasc Nurs. 2023 Apr 12;22(3):245-253. doi: 10.1093/eurjcn/zvac080. PMID 36062451
- [Derived] Koehler F, Koehler K, Prescher S, Kirwan BA, Wegscheider K, Vettorazzi E, Lezius S, Winkler S, Moeller V, Fiss G, Schleder J, Koehler M, Zugck C, Stork S, Butter C, Prondzinsky R, Spethmann S, Angermann C, Stangl V, Halle M, von Haehling S, Dreger H, Stangl K, Deckwart O, Anker SD. Mortality and morbidity 1 year after stopping a remote patient management intervention: extended follow-up results from the telemedical interventional management in patients with heart failure II (TIM-HF2) randomised trial. Lancet Digit Health. 2020 Jan;2(1):e16-e24. doi: 10.1016/S2589-7500(19)30195-5. Epub 2019 Dec 12. PMID 33328035
- [Derived] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Winkler S, Vettorazzi E, Polze A, Stangl K, Hartmann O, Marx A, Neuhaus P, Scherf M, Kirwan BA, Anker SD. Telemedical Interventional Management in Heart Failure II (TIM-HF2), a randomised, controlled trial investigating the impact of telemedicine on unplanned cardiovascular hospitalisations and mortality in heart failure patients: study design and description of the intervention. Eur J Heart Fail. 2018 Oct;20(10):1485-1493. doi: 10.1002/ejhf.1300. Epub 2018 Sep 19. PMID 30230666
- [Derived] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Kirwan BA, Winkler S, Vettorazzi E, Bruch L, Oeff M, Zugck C, Doerr G, Naegele H, Stork S, Butter C, Sechtem U, Angermann C, Gola G, Prondzinsky R, Edelmann F, Spethmann S, Schellong SM, Schulze PC, Bauersachs J, Wellge B, Schoebel C, Tajsic M, Dreger H, Anker SD, Stangl K. Efficacy of telemedical interventional management in patients with heart failure (TIM-HF2): a randomised, controlled, parallel-group, unmasked trial. Lancet. 2018 Sep 22;392(10152):1047-1057. doi: 10.1016/S0140-6736(18)31880-4. Epub 2018 Aug 25. PMID 30153985
- See also: study website, only in German — http://www.fontane-studie.de
- See also: project website, only in German — http://www.gesundheitsregion-fontane.de